CLINICAL TRIAL: NCT06779266
Title: Endoscopic Hand Suturing in the Prevention of Gastrointestinal Bleeding After Gastric Endoscopic Submucosal Dissection.
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Zofia Orzeszko, Principal Investigator, Jagiellonian University
Other Study IDs: 2025-0101
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Endoscopic Surgical Procedures
Keywords: Endoscopic Hand Suturing; Suturing Techniques; Endoscopic Submucosal Dissection; Gastrointestinal Bleeding; Endoscopic Closure Techniques
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Sutures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No closure: Participants who underwent endoscopic submucosal dissection without additional closure of the resection site.
  Interventions: Procedure: No closure
- Sutured: Participants who underwent endoscopic submucosal dissection followed by closure of the resection site with through-the-scope suturing.
  Interventions: Procedure: Suturing
- Clipped: Participants who underwent endoscopic submucosal dissection followed by closure of the resection site with through-the-scope clips.
  Interventions: Procedure: Clipping

INTERVENTIONS:
Procedure: Suturing — Endoscopic Suturing is a technique of the wound closure after advanced endoscopic third-space resections in the upper and lower gastrointestinal tract. In this technique, the needle is held on the opposite side from the tip with the needle holder. The needle is pierced perpendicularly into the tissue at the side of the wound with an appropriate margin, then driven through the tissue with rotation and grasped at the bottom of the defect. The same steps are repeated from the middle of the wound to create a symmetrical structure.
  Other Names: Endoscopic Hand Suturing; Endoscopic Through-the-scope Suturing
  Groups: Sutured
Procedure: Clipping — Clipping is a technique of the wound closure after advanced endoscopic third-space resections I the upper and lower gastrointestinal tract. In this technique, the through-the-scope clips are delivered to the site through the working canal. The arms of the clip are properly put on the both sides of the defect and the clip is closed to seal the margins. The procedure may be repeated along the resection site for complete closure.
  Other Names: Endoscopic Through-the-scope Suturing
  Groups: Clipped
Procedure: No closure — The resection site after endoscopic submucosal dissection was left open, without additional closure.
  Groups: No closure

SUMMARY:
Endoscopic hand-suturing (EHS) is a significant improvement in gastrointestinal advanced endoscopic procedures. Evidence supporting its effectiveness in clinical practice is limited due to its recent introduction and limited availability. This study aims to demonstrate the feasibility of EHS following advanced endoscopic submucosal dissection (ESD) in the stomach and investigate its potential to prevent gastrointestinal bleeding.

DETAILED DESCRIPTION:
Endoscopic hand-suturing (EHS) is a significant improvement in gastrointestinal advanced endoscopic procedures. Evidence supporting its effectiveness in clinical practice is limited due to its recent introduction and limited availability. This study aims to demonstrate the feasibility of EHS following advanced endoscopic submucosal dissection (ESD) in the stomach and investigate its potential to prevent gastrointestinal bleeding. The retrospective single-center study included individuals who underwent endoscopic submucosal dissection in the stomach. The resection site was either left open, clipped, or sutured. The study evaluated the overall procedure time (OPT), bleeding rate (BR), perforation rate, and length of hospital stay (HS). The assessment was conducted to compare the outcomes of "non-sutured vs. sutured" "no closure vs. closure" and "clipped vs. sutured" along with the propensity score matching analysis for reducing a potential selection bias.

ELIGIBILITY:
Inclusion Criteria:

* underwent gastric ESD from June 2015 to June 2024
* Eastern Cooperative Oncology Group performance status score of 0 or 1

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective study included all individuals who underwent gastric ESD from June 2015 to June 2024 in a single high-volume center and had an Eastern Cooperative Oncology Group performance status score of 0 or 1. All included procedures were performed in a conventional manner. The resection site was either left open, clipped, or sutured.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Delayed bleeding (DB) rate | 28 days
  symptomatic bleeding occurring after the ESD procedure and within 28 days following the treatment. The symptoms included hematemesis, melena, and decrease in hemoglobin >2g/dL.

SECONDARY OUTCOMES:
Overall Procedure Time (OPT) | procedural
  Measured in minutes and based on the procedural protocol.
Perforation Rate | 28 days
  Defined as post-procedural clinical signs of peritonitis with radiological signs of air in the peritoneal cavity.
Length of Hospital Stay (HS) | 28 days
  The time from the procedure to the discharge measured in days and based on the hospital database.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Spychalski, Prof., Study Chair — Medical University of Lodz; Zofia Orzeszko, MD, Principal Investigator — Jagiellonian University in Cracow
Locations (1):
- Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We intend to share the encrypted data with other investigators after appropriate application and approval of the study chair.

REFERENCES:
- [Background] Jiang W, Cen L, Dong C, Zhu S, Shen Z, Li D. Prophylactic Clipping to Prevent Delayed Bleeding and Perforation After Endoscopic Submucosal Dissection and Endoscopic Mucosal Resection: A Systematic Review and Meta-analysis. J Clin Gastroenterol. 2022 Sep 1;56(8):643-653. doi: 10.1097/MCG.0000000000001721. Epub 2022 May 25. PMID 35648969
- [Background] Goto O, Morita Y, Takayama H, Hirasawa K, Sato C, Oyama T, Takahashi A, Abe S, Saito Y, Ono H, Kawata N, Otsuka T, Iwakiri K. Endoscopic hand suturing has the potential to reduce bleeding after gastric endoscopic submucosal dissection in patients on antithrombotic agents: Multicenter phase II study. Dig Endosc. 2025 Mar;37(3):266-274. doi: 10.1111/den.14911. Epub 2024 Aug 28. PMID 39193787
- [Background] Jia Y, Zhai G, Wang E, Li P. Efficacy of local hemostatic agents after endoscopic submucosal dissection: a meta-analysis. Minim Invasive Ther Allied Technol. 2022 Oct;31(7):1017-1025. doi: 10.1080/13645706.2022.2111217. Epub 2022 Aug 24. PMID 36000962
- [Background] Libanio D, Pimentel-Nunes P, Bastiaansen B, Bisschops R, Bourke MJ, Deprez PH, Esposito G, Lemmers A, Leclercq P, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, Fuccio L, Bhandari P, Dinis-Ribeiro M. Endoscopic submucosal dissection techniques and technology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review. Endoscopy. 2023 Apr;55(4):361-389. doi: 10.1055/a-2031-0874. Epub 2023 Mar 7. PMID 36882090
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503